CLINICAL TRIAL: NCT06433492
Title: Safety and Efficacy of Viscosupplementation of Hyaluronic Acid With Addition of Liposomes in Patients With Mild or Moderate Osteoarthrosis of the Knee Joint.
Brief Title: Safety and Efficacy of Viscosupplementation of Hyaluronic Acid With Addition of Lecithin in Patients With Mild or Moderate Osteoarthrosis of the Knee Joint.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biovico Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.0 06.10.2020
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections, Intra-Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): 50 patients age 38-70 with OA confirmed by ACR criteria and radiologically verified OA (Kellgren-Lawrence grade 2 or 3) suffering from knee joint pain for at least 3 months and VAS pain score minimum 4 in one knee, and < 2 in the contralateral knee were subjected to the administration of Lipotris™. The product was administered as a course of three injections weekly.
  Interventions: Device: Intra-articular injection

INTERVENTIONS:
Device: Intra-articular injection — Three doses of intra-articular injection administered in weekely intervals.

SUMMARY:
The main objective of this prospective, open-label clinical trial is to assess the effectiveness and safety of intra-articular liposomal gel therapy for knee OA symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 38 and 70 years,
* OA diagnosed by the American College of Rheumatology (ACR) criteria,
* OA diagnosed by radiographic imaging (grade II - III according to the Kellgren-Lawrence scale),
* Pain in the knee joint for at least 3 months,
* Screening pain intensity in the target knee measured on VAS scale was required to be 4 for symptomatic knee and 2 for the contralateral knee.

Exclusion Criteria:

* Previous injections of hyaluronic acid or platelet-rich plasma within 6 months or corticosteroid injections within 3 months before the enrollment,
* Present joint infection,
* Previous knee arthroscopy up to 1 year prior to examination,
* Peripheral inflammatory and autoimmune diseases that progress with joint involvement (rheumatoid arthritis, spondyloarthropathies, systemic lupus erythematosus etc.),
* Total arthroplasty and osteotomy,
* Ankylosis of the study joint,
* Dermatitis or dermatological disease at the intended injection site,
* Known hypersensitivity to the components of the preparation,
* Coexistence of the degenerative changes in other limb joints (hip, foot),
* Cancer,
* Oral corticosteroid therapy,
* Use of medicines that affect blood clotting (heparins, oral anticoagulants, thrombolytic drugs),
* Pregnancy or breast-feeding.
* History of injury to the knee, a broken bone or dislocation of a joint, other musculoskeletal diseases that affect the study joint, neoplastic disease.
* Participation in other clinical trials.

Ages: 38 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
The pain score of Visual Analog Scale (VAS) of target knee at 3 months post-treatment. | 3 months
  The visual analog scale (VAS) measures the severity of pain. The patient assesses the level of pain by marking a point on a line 10 cm long, where a value of 0 is assigned the complete absence of pain, and a value of 10 is assigned the most severe pain the patient can imagine.

SECONDARY OUTCOMES:
The pain score of VAS of target knee at baseline, 1 week, 2 weeks, 1 month, and 6 months post-treatment | baseline, 1 week, 2 weeks, 1 month, and 6 months post-treatment
  The pain score of VAS of target knee at baseline, 1 week, 2 weeks, 1 month, and 6 months post-treatment.
The score of WOMAC at baseline, 1 week, 2 weeks, 1 month, 3 months and 6 months post-treatment | baseline, 1 week, 2 weeks, 1 month, 3 months and 6 months post-treatment
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of hip and knee osteoarthritis. It is a self-administered questionnaire consisting of 24 items.The patient assesses his condition using a scale by marking one of 5 options (scoring 0 - 4, where 0 - no complaints, 1 - mild, 2 - moderate, 3 - severe, 4 - extreme). The scores for each subscale are summed up to give a total subscale score, with higher scores indicating greater severity of symptoms.
Functional status of knee joint according to time to perform the The Timed Up and Go Test. | baseline, 1 month, 3 months and 6 months post-treatment
  The TUG test measures the time it takes for a person to stand up from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Functional status of knee joint according to time to perform the Five Time Sit to Stand Test. | baseline, 1 month, 3 months and 6 months post-treatment
  To perform "The Five Time Sit to Stand Test" (FTSST, 5xSTS), patient was asked to take a sitting position on a standard 45 cm high chair with arms crossed over the chest. At the command "START," the patient must stand up as quickly as possible five times and completely straighten up and sit back in the chair without supporting himself with his arms.
Functional status of knee joint according to time to perform the to 10 Meter Walk Test. | baseline, 1 month, 3 months and 6 months post-treatment
  The 10 Meter Walk Test (10MWT) is a clinical assessment tool used to evaluate a patient's walking speed and mobility. The test involves measuring the time it takes for a patient to walk 10 meters (33 feet) at normal, self-selected pace.
Maximum isometric force of flexor muscles of knee joint. | baseline, 1 month, 3 months and 6 months post-treatment
  Maximal voluntary isometric contraction (MVIC) of extensor/flexor muscles of knee joint measurement was performed with Forcemeter FB 500 (AXIS, Gdansk, Poland). To measure the maximum isometric force of the knee joint extensors/flexors, a person sits on a bench with the belt around waist and legs placed freely beyond the table. The measuring belt is placed parallel to the floor just above the ankle joint with knee flexed to 90 degrees. The length of the measuring belt is specified 160 cm for extensors and 60 cm for flexors. The procedure starts with the measuring belt pretension, then the patient is asked to extend/flex the knee as hard as patient can and hold it for 6 s.
Maximum isometric force of extensor muscles of the knee joint. | baseline, 1 month, 3 months and 6 months post-treatment
Safety assesment | baseline, 1 month, 3 months and 6 months post-treatment
  Number of patients with adverse events -type, duration and severity of every adverse event for each patient will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Rehasport, Poznan, Poland